CLINICAL TRIAL: NCT00904449
Title: An Open-Label Assessment of the Long-Term Safety and Utility of Numorphan® for the Relief of Moderate to Severe Pain in Patients With Cancer
Brief Title: Open Label Assessment of Long-Term Safety and Utility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director Clinical R&D, Endo Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3202-022
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: Oxymorphone ER

INTERVENTIONS:
Drug: Oxymorphone ER — 10mg, 20mg, and 40mg PO

SUMMARY:
The purpose of this study is to monitor the long-term analgesic effectiveness, safety, and utility of oxymorphone ER for the relief of moderate to severe pain due to cancer.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged > 18 years with moderate to severe pain arising from cancer (histologically and/or clinically proven) who require chronic treatment with WHO step 3 analgesics.
* Women of child-bearing potential must be using an approved method of contraception (hormone contraception, IUD, or double barrier method) and have a negative serum pregnancy test prior to entry into the study.
* Participated in study EN3202-018; the patient must have been treated with study medication and completed the exit visit to be eligible.

Exclusion Criteria:

* Experienced a serious, adverse experience during study EN3202-018 that was possible or probably related to study medication.
* Withdrew from study EN3202-018 due to an Adverse experience possibly or probably related to study medication.
* Known idiosyncratic reaction or hypersensitivity to oxymorphone.
* Inability to take oral medication for 1 week.
* Patients with ileosomy, mechanical intestinal obstruction, partial or complete gastric outlet obstruction, parlayticileus, or other conditions that might contraindicate the use of, or impair the absorption of an oral controlled-release dosage form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-04; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Assessment of AEs and clinical laboratory values | 22 months

SECONDARY OUTCOMES:
Favorable long-term safety profile for oxymorhpone ER in the treatment of moderate to severe pain in patients with cancer | 22 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals